CLINICAL TRIAL: NCT05560971
Title: The Effect of Palmitoleic Acid (POA) Supplementation on Insulin Sensitivity and Lipogenesis in Overweight and Obese Individuals
Brief Title: Monounsaturated Fatty Acid Supplementation for Overweight and Obese Individuals With Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Tersus Life Sciences LLC (Industry)
Responsible Party: Principal Investigator, Mehmet F. Burak, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022P001764
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: PreDiabetes; Insulin Resistance; Overweight; Obesity
Keywords: Palmitoleic acid; Obesity; Insulin resistance; Dietary supplement; Prediabetes
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Overweight; Obesity | interventions — palmitoleic acid

STUDY DESIGN:
Intervention Model Description: Interventional double-blinded study with participants randomized to either POA or placebo
Who Masked: Participant, Investigator
Masking Description: Participants and study staff both blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palmitoleic acid (Active Comparator): The treatment arm will receive Palmitoleic acid (POA) supplement as Provinal® 420 mg capsules with at least 90% pure POA Ethyl Ester (less than 1% palmitic acid). Participants will be asked to consume 2 Provinal® 420 mg capsules twice a day for 8 weeks.
  Interventions: Dietary Supplement: Palmitoleic acid
- Placebo (Placebo Comparator): The placebo is a medium chain fatty acid in triglyceride form. The placebo has no shown health effects, neither beneficial or detrimental. Participants will be asked to consume 2 placebo capsules daily twice a day for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Palmitoleic acid — Participants will be randomized to either POA or placebo and will be asked to take 2 capsules of the POA or placebo twice a day for 8 weeks.
  Other Names: Provinal®
  Arms: Palmitoleic acid
Other: Placebo — Medium chain fatty acids in triglyceride form in capsules with the same shape, color, size and odor of POA capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand and determine whether Palmitoleic acid (POA), monounsaturated omega-7 fatty acid (exists in regular diet), improves insulin sensitivity and decreases liver fat accumulation in humans. Unlike others, the study will use POA as a dietary supplement, rather than complex oils, which contain a significant amount of saturated fat palmitic acid. Palmitic acid has known harmful effects on the body. Hence, eliminating palmitic acid from supplementation of POA might increase its benefits. This trial stems from the preclinical discoveries that POA acting as a fat hormone, has beneficial effects on the liver, muscle, vessels, and fat tissue. Supporting this, higher POA levels in humans have been shown to be correlated with a reduced risk of developing type-2 diabetes and cardiovascular diseases such as heart attacks. In animals, it has been observed that POA improves sugar metabolism in a number of mechanisms related to the liver and muscle. Based on these findings, the design of this study is a double-blind placebo-controlled trial that tests the effects of POA on insulin sensitivity of overweight and obese adult individuals with pre-diabetes.

DETAILED DESCRIPTION:
Specific aims of the study are as follows: 1) To test whether supplementation of POA, as compared to placebo, improves insulin sensitivity. 2) To test whether supplementation of POA, as compared to placebo, ameliorates hepatosteatosis and decreases whole-body fat mass, serum triglyceride, and LDL cholesterol. 3)To determine whether supplementation of POA, as compared to placebo, decreases plasma levels of fasting glucose, insulin, FABP4, glucagon, inflammatory cytokines, and hsCRP.

The investigators will recruit overweight and obese individuals (BMI 25-40) with mild insulin resistance, prediabetes and/or impaired glucose tolerance. The study is powered only for the primary endpoint, insulin sensitivity. After the screening visit confirms the eligibility for the study; the investigators will perform an oral glucose tolerance test (OGTT) for stratified randomization for better homogeneity between POA and placebo groups. The investigators aim to have 40 participants complete the study which will consist of 2 main overnight visits consisting of an insulin clamp procedure and a mixed meal tolerance test the night prior. Participants will also have a liver MRI and DEXA scan at these two visits. Participants will be asked to consume a palmitoleic acid minimized diet for 10 weeks which will start two weeks before the first overnight visit. This research study will compare insulin sensitivity before and 8 weeks after taking POA vs placebo in the same individuals. After the first overnight visit participants will be given either POA or placebo capsules to take daily for 8 weeks until the second overnight visit. There will also be a short blood draw visit 4 weeks after the first overnight visit.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese individuals with prediabetes and/or impaired glucose tolerance
* Age 18 to 70 years
* BMI 25-40 kg/m2
* HbA1c between 5.6 - 6.5, Impaired fasting plasma glucose levels (>99, ≤126 mg/dL) or OGTT blood glucose at 2 hours between 140-200 mg/dL or HOMA-IR >2.5
* BP <150/90 with or without medication
* GFR>60
* ALT, AST <300
* Normal thyroid function is defined as screening TSH within normal ranges, with or without medication

Exclusion Criteria:

* Use of any medications (except thyroid hormone with normal TSH, anti-hypertensives with blood pressure <150/90 and non-steroidal rescue inhalers for asthma)
* Pregnancy or breastfeeding
* Use of over-the-counter (OTC) supplements (except vitamin D). The investigators will ensure that study participants are not using supplements containing fish oil or other lipid supplements (e.g., macadamia oil, krill oil, flaxseed, primrose oil, sea buckthorn oil) within 3 months of study participation
* Greater than 3 servings/day combined of cheese, whole-fat milk, kefir, or whole-fat yogurt for the last 3 months before the study.
* Diagnosed with any type of diabetes mellitus and/or taking glucose-lowering medications
* Recent weight loss (more than 7% of total body weight loss in last 3 months)
* Established major chronic diseases such as major cardiovascular disease (history of myocardial infarction, stroke, symptomatic heart failure, coronary artery bypass graft, Atrial fibrillation, symptomatic peripheral arterial disease), bleeding disorder or anticoagulation use, active cancer, end-stage renal disease, proteinuria (>3g/day), dementia, severe chronic obstructive pulmonary disease (needs systemic steroid therapy), significant liver disease (ALT or AST>300)
* History of ongoing smoking cigarettes >1 pack/day, alcohol abuse, or illicit drug abuse
* Treatment with any investigational drug in the one month preceding the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity M value change before and 8 weeks after POA vs placebo intake | 8 weeks
  Insulin sensitivity (M values) will be evaluated by hyperinsulinemic euglycemic clamp (gold standard) from the same individuals before and after taking POA vs. placebo. The investigators will compare M values before and after taking POA vs placebo intake. Hence the investigators are looking for delta changes and expect 20% statistically significant improvement with POA and no significant change with placebo. The investigators calculated sample size and powered the study for only this primary endpoint to see at least 20% difference.

SECONDARY OUTCOMES:
Modified mixed meal tolerance test | 8 weeks
  The investigators will measure glucose and c-peptide response to standard mixed meal. Study participants will ingest the mixed meal and then the investigators will measure glucose and c-peptide levels from venous blood collected every 30 minutes for 2 hours. Area under the curve (AUC) for both glucose and c-peptide will be calculated and this value from same individuals before and 8 weeks after POA vs placebo intake will be compared.
Liver fat quantification | 8 weeks
  Liver fat percent will be evaluated by liver MRI-PDFF (proton density fat fraction). Blinded radiologist will analyze the MRI fat fraction and use standard ROI gating. The investigators will compare % fat fraction (FF) from same individuals before and 8 weeks after POA vs placebo intake
Total body fat mass and body composition | 8 weeks
  Body composition, which is whole-body fat vs lean mass will be evaluated by DEXA scan. Whole-body % fat mass from same individuals before and 8 weeks after POA vs placebo intake will be compared.
Serum; fasting glucose, insulin, LDL cholesterol, hsCRP, circulating inflammatory cytokines (TNF-a, IL-6), FABP4, glucagon | 8 weeks
  The investigoators will compare serum fasting glucose, insulin, LDL cholesterol, hsCRP, circulating inflammatory cytokines (TNF-a, IL-6), FABP4, glucagon from same individuals before and 8 weeks after POA vs placebo intake

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Furkan Burak, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burak MF, Inouye KE, White A, Lee A, Tuncman G, Calay ES, Sekiya M, Tirosh A, Eguchi K, Birrane G, Lightwood D, Howells L, Odede G, Hailu H, West S, Garlish R, Neale H, Doyle C, Moore A, Hotamisligil GS. Development of a therapeutic monoclonal antibody that targets secreted fatty acid-binding protein aP2 to treat type 2 diabetes. Sci Transl Med. 2015 Dec 23;7(319):319ra205. doi: 10.1126/scitranslmed.aac6336. Epub 2015 Dec 23. PMID 26702093
- [Background] Cao H, Sekiya M, Ertunc ME, Burak MF, Mayers JR, White A, Inouye K, Rickey LM, Ercal BC, Furuhashi M, Tuncman G, Hotamisligil GS. Adipocyte lipid chaperone AP2 is a secreted adipokine regulating hepatic glucose production. Cell Metab. 2013 May 7;17(5):768-78. doi: 10.1016/j.cmet.2013.04.012. PMID 23663740
- [Background] Cao H, Gerhold K, Mayers JR, Wiest MM, Watkins SM, Hotamisligil GS. Identification of a lipokine, a lipid hormone linking adipose tissue to systemic metabolism. Cell. 2008 Sep 19;134(6):933-44. doi: 10.1016/j.cell.2008.07.048. PMID 18805087
- [Background] Olefsky JM. Fat talks, liver and muscle listen. Cell. 2008 Sep 19;134(6):914-6. doi: 10.1016/j.cell.2008.09.001. PMID 18805083
- [Background] Dimopoulos N, Watson M, Sakamoto K, Hundal HS. Differential effects of palmitate and palmitoleate on insulin action and glucose utilization in rat L6 skeletal muscle cells. Biochem J. 2006 Nov 1;399(3):473-81. doi: 10.1042/BJ20060244. PMID 16822230
- [Background] Maedler K, Spinas GA, Dyntar D, Moritz W, Kaiser N, Donath MY. Distinct effects of saturated and monounsaturated fatty acids on beta-cell turnover and function. Diabetes. 2001 Jan;50(1):69-76. doi: 10.2337/diabetes.50.1.69. PMID 11147797
- [Background] Maedler K, Oberholzer J, Bucher P, Spinas GA, Donath MY. Monounsaturated fatty acids prevent the deleterious effects of palmitate and high glucose on human pancreatic beta-cell turnover and function. Diabetes. 2003 Mar;52(3):726-33. doi: 10.2337/diabetes.52.3.726. PMID 12606514
- [Background] Gravena C, Mathias PC, Ashcroft SJ. Acute effects of fatty acids on insulin secretion from rat and human islets of Langerhans. J Endocrinol. 2002 Apr;173(1):73-80. doi: 10.1677/joe.0.1730073. PMID 11927386
- [Background] Cimen I, Kocaturk B, Koyuncu S, Tufanli O, Onat UI, Yildirim AD, Apaydin O, Demirsoy S, Aykut ZG, Nguyen UT, Watkins SM, Hotamisligil GS, Erbay E. Prevention of atherosclerosis by bioactive palmitoleate through suppression of organelle stress and inflammasome activation. Sci Transl Med. 2016 Sep 28;8(358):358ra126. doi: 10.1126/scitranslmed.aaf9087. PMID 27683551
- [Background] Duckett SK, Volpi-Lagreca G, Alende M, Long NM. Palmitoleic acid reduces intramuscular lipid and restores insulin sensitivity in obese sheep. Diabetes Metab Syndr Obes. 2014 Nov 20;7:553-63. doi: 10.2147/DMSO.S72695. eCollection 2014. PMID 25429233
- [Background] Yang ZH, Miyahara H, Hatanaka A. Chronic administration of palmitoleic acid reduces insulin resistance and hepatic lipid accumulation in KK-Ay Mice with genetic type 2 diabetes. Lipids Health Dis. 2011 Jul 21;10:120. doi: 10.1186/1476-511X-10-120. PMID 21774832
- [Background] Lima EA, Silveira LS, Masi LN, Crisma AR, Davanso MR, Souza GI, Santamarina AB, Moreira RG, Martins AR, de Sousa LG, Hirabara SM, Rosa Neto JC. Macadamia oil supplementation attenuates inflammation and adipocyte hypertrophy in obese mice. Mediators Inflamm. 2014;2014:870634. doi: 10.1155/2014/870634. Epub 2014 Sep 22. PMID 25332517
- [Background] Riserus U, Willett WC, Hu FB. Dietary fats and prevention of type 2 diabetes. Prog Lipid Res. 2009 Jan;48(1):44-51. doi: 10.1016/j.plipres.2008.10.002. Epub 2008 Nov 7. PMID 19032965
- [Background] Guo X, Jiang X, Chen K, Liang Q, Zhang S, Zheng J, Ma X, Jiang H, Wu H, Tong Q. The Role of Palmitoleic Acid in Regulating Hepatic Gluconeogenesis through SIRT3 in Obese Mice. Nutrients. 2022 Apr 1;14(7):1482. doi: 10.3390/nu14071482. PMID 35406095
- [Background] Bolsoni-Lopes A, Festuccia WT, Chimin P, Farias TS, Torres-Leal FL, Cruz MM, Andrade PB, Hirabara SM, Lima FB, Alonso-Vale MI. Palmitoleic acid (n-7) increases white adipocytes GLUT4 content and glucose uptake in association with AMPK activation. Lipids Health Dis. 2014 Dec 20;13:199. doi: 10.1186/1476-511X-13-199. PMID 25528561
- [Background] de Souza CO, Teixeira AAS, Biondo LA, Lima Junior EA, Batatinha HAP, Rosa Neto JC. Palmitoleic Acid Improves Metabolic Functions in Fatty Liver by PPARalpha-Dependent AMPK Activation. J Cell Physiol. 2017 Aug;232(8):2168-2177. doi: 10.1002/jcp.25715. Epub 2017 Mar 24. PMID 27925195
- [Background] Yang ZH, Takeo J, Katayama M. Oral administration of omega-7 palmitoleic acid induces satiety and the release of appetite-related hormones in male rats. Appetite. 2013 Jun;65:1-7. doi: 10.1016/j.appet.2013.01.009. Epub 2013 Jan 30. PMID 23376733
- [Background] Tovar R, Gavito AL, Vargas A, Soverchia L, Hernandez-Folgado L, Jagerovic N, Baixeras E, Ciccocioppo R, Rodriguez de Fonseca F, Decara J. Palmitoleoylethanolamide Is an Efficient Anti-Obesity Endogenous Compound: Comparison with Oleylethanolamide in Diet-Induced Obesity. Nutrients. 2021 Jul 28;13(8):2589. doi: 10.3390/nu13082589. PMID 34444748
- [Background] Chan KL, Pillon NJ, Sivaloganathan DM, Costford SR, Liu Z, Theret M, Chazaud B, Klip A. Palmitoleate Reverses High Fat-induced Proinflammatory Macrophage Polarization via AMP-activated Protein Kinase (AMPK). J Biol Chem. 2015 Jul 3;290(27):16979-88. doi: 10.1074/jbc.M115.646992. Epub 2015 May 18. PMID 25987561
- [Background] de Souza CO, Valenzuela CA, Baker EJ, Miles EA, Rosa Neto JC, Calder PC. Palmitoleic Acid has Stronger Anti-Inflammatory Potential in Human Endothelial Cells Compared to Oleic and Palmitic Acids. Mol Nutr Food Res. 2018 Oct;62(20):e1800322. doi: 10.1002/mnfr.201800322. Epub 2018 Aug 28. PMID 30102465
- [Background] Weimann E, Silva MBB, Murata GM, Bortolon JR, Dermargos A, Curi R, Hatanaka E. Topical anti-inflammatory activity of palmitoleic acid improves wound healing. PLoS One. 2018 Oct 11;13(10):e0205338. doi: 10.1371/journal.pone.0205338. eCollection 2018. PMID 30307983
- [Background] Tang J, Yang B, Yan Y, Tong W, Zhou R, Zhang J, Mi J, Li D. Palmitoleic Acid Protects against Hypertension by Inhibiting NF-kappaB-Mediated Inflammation. Mol Nutr Food Res. 2021 Jun;65(12):e2001025. doi: 10.1002/mnfr.202001025. Epub 2021 May 10. PMID 33865240
- [Background] Trico D, Mengozzi A, Nesti L, Hatunic M, Gabriel Sanchez R, Konrad T, Lalic K, Lalic NM, Mari A, Natali A; EGIR-RISC Study Group. Circulating palmitoleic acid is an independent determinant of insulin sensitivity, beta cell function and glucose tolerance in non-diabetic individuals: a longitudinal analysis. Diabetologia. 2020 Jan;63(1):206-218. doi: 10.1007/s00125-019-05013-6. Epub 2019 Nov 1. PMID 31676981
- [Background] Mozaffarian D, Cao H, King IB, Lemaitre RN, Song X, Siscovick DS, Hotamisligil GS. Circulating palmitoleic acid and risk of metabolic abnormalities and new-onset diabetes. Am J Clin Nutr. 2010 Dec;92(6):1350-8. doi: 10.3945/ajcn.110.003970. Epub 2010 Oct 13. PMID 20943795
- [Background] Stefan N, Kantartzis K, Celebi N, Staiger H, Machann J, Schick F, Cegan A, Elcnerova M, Schleicher E, Fritsche A, Haring HU. Circulating palmitoleate strongly and independently predicts insulin sensitivity in humans. Diabetes Care. 2010 Feb;33(2):405-7. doi: 10.2337/dc09-0544. Epub 2009 Nov 4. PMID 19889804
- [Background] Hiraoka-Yamamoto J, Ikeda K, Negishi H, Mori M, Hirose A, Sawada S, Onobayashi Y, Kitamori K, Kitano S, Tashiro M, Miki T, Yamori Y. Serum lipid effects of a monounsaturated (palmitoleic) fatty acid-rich diet based on macadamia nuts in healthy, young Japanese women. Clin Exp Pharmacol Physiol. 2004 Dec;31 Suppl 2:S37-8. doi: 10.1111/j.1440-1681.2004.04121.x. PMID 15649284
- [Background] Garg ML, Blake RJ, Wills RB. Macadamia nut consumption lowers plasma total and LDL cholesterol levels in hypercholesterolemic men. J Nutr. 2003 Apr;133(4):1060-3. doi: 10.1093/jn/133.4.1060. PMID 12672919
- [Background] Curb JD, Wergowske G, Dobbs JC, Abbott RD, Huang B. Serum lipid effects of a high-monounsaturated fat diet based on macadamia nuts. Arch Intern Med. 2000 Apr 24;160(8):1154-8. doi: 10.1001/archinte.160.8.1154. PMID 10789609
- [Background] Griel AE, Cao Y, Bagshaw DD, Cifelli AM, Holub B, Kris-Etherton PM. A macadamia nut-rich diet reduces total and LDL-cholesterol in mildly hypercholesterolemic men and women. J Nutr. 2008 Apr;138(4):761-7. doi: 10.1093/jn/138.4.761. PMID 18356332
- [Background] Pinnick KE, Neville MJ, Fielding BA, Frayn KN, Karpe F, Hodson L. Gluteofemoral adipose tissue plays a major role in production of the lipokine palmitoleate in humans. Diabetes. 2012 Jun;61(6):1399-403. doi: 10.2337/db11-1810. Epub 2012 Apr 9. PMID 22492525
- [Background] Imamura F, Fretts A, Marklund M, Ardisson Korat AV, Yang WS, Lankinen M, Qureshi W, Helmer C, Chen TA, Wong K, Bassett JK, Murphy R, Tintle N, Yu CI, Brouwer IA, Chien KL, Frazier-Wood AC, Del Gobbo LC, Djousse L, Geleijnse JM, Giles GG, de Goede J, Gudnason V, Harris WS, Hodge A, Hu F; InterAct Consortium; Koulman A, Laakso M, Lind L, Lin HJ, McKnight B, Rajaobelina K, Riserus U, Robinson JG, Samieri C, Siscovick DS, Soedamah-Muthu SS, Sotoodehnia N, Sun Q, Tsai MY, Uusitupa M, Wagenknecht LE, Wareham NJ, Wu JH, Micha R, Forouhi NG, Lemaitre RN, Mozaffarian D; Fatty Acids and Outcomes Research Consortium (FORCE). Fatty acid biomarkers of dairy fat consumption and incidence of type 2 diabetes: A pooled analysis of prospective cohort studies. PLoS Med. 2018 Oct 10;15(10):e1002670. doi: 10.1371/journal.pmed.1002670. eCollection 2018 Oct. PMID 30303968
- [Background] Dyerberg J, Bang HO, Hjorne N. Fatty acid composition of the plasma lipids in Greenland Eskimos. Am J Clin Nutr. 1975 Sep;28(9):958-66. doi: 10.1093/ajcn/28.9.958. PMID 1163480
- [Background] Bang HO, Dyerberg J, Hjoorne N. The composition of food consumed by Greenland Eskimos. Acta Med Scand. 1976;200(1-2):69-73. doi: 10.1111/j.0954-6820.1976.tb08198.x. PMID 961471
- [Background] Adler GK, Hornik ES, Murray G, Bhandari S, Yadav Y, Heydarpour M, Basu R, Garg R, Tirosh A. Acute effects of the food preservative propionic acid on glucose metabolism in humans. BMJ Open Diabetes Res Care. 2021 Jul;9(1):e002336. doi: 10.1136/bmjdrc-2021-002336. PMID 34312159
- [Background] Kampmann U, Mosekilde L, Juhl C, Moller N, Christensen B, Rejnmark L, Wamberg L, Orskov L. Effects of 12 weeks high dose vitamin D3 treatment on insulin sensitivity, beta cell function, and metabolic markers in patients with type 2 diabetes and vitamin D insufficiency - a double-blind, randomized, placebo-controlled trial. Metabolism. 2014 Sep;63(9):1115-24. doi: 10.1016/j.metabol.2014.06.008. Epub 2014 Jun 19. PMID 25044176
- [Background] Tripathy D, Wessman Y, Gullstrom M, Tuomi T, Groop L. Importance of obtaining independent measures of insulin secretion and insulin sensitivity during the same test: results with the Botnia clamp. Diabetes Care. 2003 May;26(5):1395-401. doi: 10.2337/diacare.26.5.1395. PMID 12716795